CLINICAL TRIAL: NCT02181517
Title: A Study of Abicipar Pegol in Patients With Neovascular Age-related Macular Degeneration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 150998-003; CYPRESS (Other: Allergan)
Record Dates: First submitted 2014-07-02; First posted 2014-07-04 (Estimated); Results first posted 2016-04-05 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-04

CONDITIONS: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — abicipar pegol; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- abicipar pegol 1 mg (Experimental): Abicipar pegol 1 mg administered to the study eye by intravitreal injection at day 1, weeks 4 and 8, followed by a sham procedure at weeks 12 and 16.
  Interventions: Drug: abicipar pegol; Other: sham procedure
- abicipar pegol 2 mg (Experimental): Abicipar pegol 2 mg administered to the study eye by intravitreal injection at day 1, weeks 4 and 8, followed by a sham procedure at weeks 12 and 16.
  Interventions: Drug: abicipar pegol; Other: sham procedure
- ranibizumab 0.5 mg (Active Comparator): Ranibizumab (Lucentis®) 0.5 mg administered to the study eye by intravitreal injection every 4 weeks from day 1 through week 16.
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: abicipar pegol — Abicipar pegol administered to the study eye by intravitreal injection at day 1, weeks 4 and 8.
  Arms: abicipar pegol 1 mg; abicipar pegol 2 mg
Drug: ranibizumab — Ranibizumab (Lucentis®) 0.5 mg administered to the study eye by intravitreal injection every 4 weeks from day 1 through week 16.
  Other Names: Lucentis®
  Arms: ranibizumab 0.5 mg
Other: sham procedure — Sham procedure to the study eye at weeks 12 and 16.
  Arms: abicipar pegol 1 mg; abicipar pegol 2 mg

SUMMARY:
This is a safety and efficacy study of abicipar pegol in patients with neovascular age-related macular degeneration to establish comparability between Japanese and non-Japanese.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of wet age-related macular degeneration in at least 1 eye
* Best corrected visual acuity of 20/32 to 20/320 in the study eye and 20/200 or better in the fellow eye

Exclusion Criteria:

* Hypersensitivity, allergy, or anaphylactic reaction to iodine
* Cataract or refractive surgery within the last 3 months
* History of vitrectomy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Phoenix, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Abicipar Pegol 1 mg | Abicipar Pegol 2 mg | Ranibizumab 0.5 mg
Started | 10 | 10 | 5
Completed | 10 | 10 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abicipar Pegol 1 mg | Abicipar Pegol 2 mg | Ranibizumab 0.5 mg | Total
Number analyzed (Participants) | 10 | 10 | 5 | 25
Age, Customized [Number; unit: participants]
  ≤ 65 years | 0 | 0 | 0 | 0
  > 65 years | 10 | 10 | 5 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 4 | 20
  Male | 1 | 3 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) in the Study Eye at Week 16 Using the Early Treatment Diabetic Retinopathy Study (ETDRS) Scale
Description: BCVA is measured using an eye chart and is reported as the number of letters read correctly using the ETDRS Scale (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved.
Time Frame: Baseline, Week 16
Population: Modified Intent-to-Treat (mITT) population included all randomized and treated participants with at least 1 follow-up visit.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Abicipar Pegol 1 mg | Abicipar Pegol 2 mg | Ranibizumab 0.5 mg
Number analyzed (Participants) | 10 | 10 | 5
letters
  Baseline | 55.2 (12.97) | 59.0 (10.36) | 57.6 (17.04)
  Change from Baseline at Week 16 | 4.4 (8.96) | 10.1 (10.5) | 15.2 (6.72)

2. Secondary Outcome: Change From Baseline in BCVA in the Study Eye at Week 20 Using the ETDRS Scale
Description: as for outcome 1
Time Frame: Baseline, Week 20
Population: mITT population included all randomized and treated participants with at least 1 follow-up visit.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Abicipar Pegol 1 mg | Abicipar Pegol 2 mg | Ranibizumab 0.5 mg
Number analyzed (Participants) | 10 | 10 | 5
letters
  Baseline | 55.2 (12.97) | 59.0 (10.36) | 57.6 (17.04)
  Change from Baseline at Week 20 | 5.6 (12.12) | 6.7 (15.98) | 14.4 (7.89)

3. Secondary Outcome: Percentage of Patients With a BCVA Gain of 15 or More Letters in the Study Eye Using the ETDRS Scale
Description: as for outcome 1
Time Frame: Baseline, Week 20
Population: mITT population included all randomized and treated participants with at least 1 follow-up visit.
Measure: Number; unit: percentage of participants
Arm/Group | Abicipar Pegol 1 mg | Abicipar Pegol 2 mg | Ranibizumab 0.5 mg
Number analyzed (Participants) | 10 | 10 | 5
percentage of participants | 30.0 | 30.0 | 60.0

4. Secondary Outcome: Percentage of Patients With a BCVA Gain of 10 or More Letters in the Study Eye Using the ETDRS Scale
Description: as for outcome 1
Time Frame: Baseline, Week 20
Population: mITT population included all randomized and treated participants with at least 1 follow-up visit.
Measure: Number; unit: percentage of participants
Arm/Group | Abicipar Pegol 1 mg | Abicipar Pegol 2 mg | Ranibizumab 0.5 mg
Number analyzed (Participants) | 10 | 10 | 5
percentage of participants | 40.0 | 40.0 | 60.0

5. Secondary Outcome: Change From Baseline in Central Retinal Thickness (CRT) in the Study Eye
Description: CRT was assessed using spectral domain optical coherence tomography (SD-OCT), a non-invasive diagnostic system providing high-resolution imaging sections of the retina. SD-OCT was performed in the study eye after pupil dilation. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 16, Week 20
Population: mITT population included all randomized and treated participants with at least 1 follow-up visit.
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Abicipar Pegol 1 mg | Abicipar Pegol 2 mg | Ranibizumab 0.5 mg
Number analyzed (Participants) | 10 | 10 | 5
microns
  Baseline | 443.8 (107.32) | 383.8 (146.90) | 348.8 (33.26)
  Change from Baseline at Week 16 | -106.5 (128.50) | -112.8 (169.75) | -124.4 (49.51)
  Change from Baseline at Week 20 | -78.2 (104.73) | -90.3 (178.22) | -110.4 (45.87)

ADVERSE EVENTS:
Arm/Group | Abicipar Pegol 1 mg | Abicipar Pegol 2 mg | Ranibizumab 0.5 mg
Serious Adverse Events (participants affected / at risk) | 1/10 | 1/10 | 0/5
Other Adverse Events (participants affected / at risk) | 5/10 | 6/10 | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abicipar Pegol 1 mg (N=10) | Abicipar Pegol 2 mg (N=10) | Ranibizumab 0.5 mg (N=5)
Pneumonia (Infections and infestations) | 0 | 1 | 0
Escherichia bacteremia (Infections and infestations) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abicipar Pegol 1 mg (N=10) | Abicipar Pegol 2 mg (N=10) | Ranibizumab 0.5 mg (N=5)
Dry eye (Eye disorders) | 1 | 1 | 0
Eye pain (Eye disorders) | 0 | 1 | 1
Oedema peripheral (General disorders) | 0 | 1 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0
Retinal vein occlusion (Eye disorders) | 0 | 1 | 0
Uveitis (Eye disorders) | 0 | 1 | 0
Vitritis (Eye disorders) | 0 | 1 | 0
Iridocyclitis (Eye disorders) | 1 | 0 | 0
Punctate keratitis (Eye disorders) | 1 | 0 | 0
Retinal haemorrhage (Eye disorders) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Visual acuity reduced (Eye disorders) | 1 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.